CLINICAL TRIAL: NCT04673877
Title: Tissue Concentrations of Vancomycin Achieved With Bier Block Administration Versus Intravenous Prophylaxis in Upper Extremity Surgery: A Randomized Controlled Trial
Brief Title: Vancomycin Tissue Concentrations by Bier Block or Intravenous Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kevin J. Renfree, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-007132
Record Dates: First submitted 2020-10-26; First posted 2020-12-17 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Infection; Hand Injury Wrist; Hand Injuries; Hand Injuries and Disorders; Hand Arthritis
MeSH Terms: conditions — Infections; Hand Injuries; Disease | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bier Block Group (Experimental): Subjects will receive antibiotic Vancomycin from a Bier Block (injected into an arm vein with a tourniquet up to keep antibiotics in the arm). Samples will be collected from bone and tissue that is normally removed during surgery.
  Interventions: Procedure: Bier Block; Drug: Vancomycin
- Systemic Intravenous IV Group (Active Comparator): Subjects will receive antibiotic Vancomycin through intravenous administration. Samples will be collected from bone and tissue that is normally removed during during surgery.
  Interventions: Drug: Systemic IV Vancomycin

INTERVENTIONS:
Drug: Systemic IV Vancomycin — 1 g of vancomycin will be delivered intravenously over a period of one hour prior to tourniquet inflation.
  Arms: Systemic Intravenous IV Group
Procedure: Bier Block — After exsanguination of the limb and elevation of the tourniquet in the prepped and draped patient, Vancomycin will be injected into a superficial vein in the hand, wrist or forearm.
  Arms: Bier Block Group
Drug: Vancomycin — 500 mg diluted in 50 cc normal saline of injection into superficial vein in the hand, wrist or forearm
  Arms: Bier Block Group

SUMMARY:
The purpose of this study is to determine whether or not giving a lower dose of antibiotics (Vancomycin) in the area where it is needed (upper extremity) is more effective at preventing infection than the current standard dose which is given intravenously (IV).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing upper extremity reconstruction by a single surgeon.
* Surgical cases will include:

  * Trapeziectomy/suspensionplasty.
  * PIPJ/MPJ arthroplasty.
  * Proximal row carpectomy.
  * Distal ulnar resection.
  * Distal radius fracture fixation.

Exclusion Criteria:

* Inability to adequately cannulate a superficial vein in the upper extremity within 5 minutes of tourniquet inflation.
* Evidence of subcutaneous extravasation in Bier block group.
* History of renal dysfunction.
* Vancomycin allergy.
* ASA>/= 3.
* History of lung cancer.
* Known HIV infection.
* History of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Tissue concentrations of vancomycin | Approximately 45-60 minutes after skin incision
  Tissue concentrations of vancomycin in the hand and wrist following Bier Block administration versus systemic IV administration

SECONDARY OUTCOMES:
Adverse Events | 1 year
  Number of adverse events reported for Bier Block administered vancomycin

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Renfree, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT04673877/Prot_SAP_000.pdf